CLINICAL TRIAL: NCT04679311
Title: High Angiotensin Converting Enzyme Activity-containing Plasma for the Treatment of Angiotensin Converting Enzyme Inhibitor-induced Angioedema
Brief Title: Treatment of Angiotensin Converting Enzyme Inhibitor-induced Angioedema
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: End of funding period
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202002126
Record Dates: First submitted 2020-12-15; First posted 2020-12-22 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Angioedema Caused by Angiotensin-Converting-Enzyme Inhibitor
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The laboratory that performs the assays and the assessor of the angioedema will be blinded to the treatment the subject received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High ACE Activity Fresh Frozen Plasma (Experimental): Subjects will be treated with 2 units of fresh frozen plasma that have been preselected to contain ACE activity ≥50 U/L
  Interventions: Biological: High ACE Activity Fresh Frozen Plasma
- Normal Saline (Placebo Comparator): Subjects will be treated with normal saline 500 cc.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: High ACE Activity Fresh Frozen Plasma — Subjects will be treated with fresh frozen plasma that has been preselected for ACE activity content of ≥ 50 U/L
  Arms: High ACE Activity Fresh Frozen Plasma
Other: Normal Saline — Subjects will be treated with normal saline 500 cc
  Arms: Normal Saline

SUMMARY:
Angiotensin Converting Enzyme (ACE) inhibitors are among the most important and widely prescribed drugs. They reduce the morbidity and mortality associated with high blood pressure, heart disease, and kidney disease. Unfortunately, their use carries the risk of causing life-threatening airway swelling in some patients. There is currently no treatment for this condition. A novel treatment approach that may reduce or completely reverse the swelling will be tested.

DETAILED DESCRIPTION:
The investigators will test the hypothesis that treatment with fresh frozen plasma that contains high levels of ACE activity will increase serum ACE activity and thereby cause the degradation of mediators of ACE inhibitor-induced angioedema, such as bradykinin and substance P, resulting in a shortening of the course of ACE inhibitor-induced angioedema.

16 patients with ACE inhibitor-induced angioedema will be randomized 1:1 to treatment with either 2 units of fresh frozen plasma that has been preselected for high ACE activity content (≥50 U/L) or an equal volume of normal saline. A baseline assessment of the severity of the angioedema will be performed and baseline serum levels of ACE activity will be determined. The severity of angioedema will be assessed and serum levels of ACE activity will be determined at specific intervals after each subject is treated.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older
* Must currently be on ACE inhibitor therapy and have received a dose within 36 hours
* Presenting with moderate to severe angioedema affecting the upper aerodigestive tract (face, lips, cheeks, tongue, soft palate/uvula, pharynx, and larynx). The severity of the angioedema attack will be determined by the subject's worst severity rating at baseline among 4 clinical domains (difficulty breathing, difficulty swallowing, voice changes, and tongue swelling) based on a clinically validated angioedema severity scale29 (Table)
* Presenting with ACE inhibitor-induced angioedema within 12 hours after onset
* All females must have a locally obtained negative pregnancy test prior to administration of the study drug. Those who have had a total hysterectomy, bilateral oophorectomy, or are two years post-menopausal do not require a pregnancy test.
* Must be able to provide written informed consent to participate in the study to fulfill all study requirements

Exclusion Criteria:

* Pregnancy and/or breast feeding
* Patients with angioedema that is likely due to causes other than ACE inhibitors, including hereditary angioedema, acquired angioedema, and allergic angioedema (food, insect bite or sting with clear response to anti-allergy medications)
* Patients exhibiting acute urticaria
* Evident clinical response to glucocorticoids, antihistamines, or epinephrine
* A family history of recurrent angioedema
* Documented intolerance to plasma
* Documented congenital deficiency of immunoglobulin A in the presence of anti-immunoglobulin A antibodies
* Patients with heart failure of the severity that precludes safe transfusion of High ACE activity plasma
* Patients with acute pulmonary edema
* Patients with morbid obesity as defined by BMI>40; morbidly obese patients have a higher volume of blood needing higher amounts of plasma and therefore will be excluded from this pilot study
* Opinion of the investigator that the patient would not be a good candidate
* Participation in a clinical study in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Weintraub, M.D., Principal Investigator — Washington University School of Medicine and the St. Louis VA Medical Center
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen SX, Hermelin D, Weintraub SJ. Possible donor-dependent differences in efficacy of fresh frozen plasma for treatment of ACE inhibitor-induced angioedema. J Allergy Clin Immunol Pract. 2019 Jul-Aug;7(6):2087-2088. doi: 10.1016/j.jaip.2019.02.027. Epub 2019 Mar 2. No abstract available. PMID 30836229

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High ACE Activity Fresh Frozen Plasma | Normal Saline
Started | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: No patients were randomized to the High ACE FFP. Study was terminated due to end of funding period.
Groups:
- Total: Total of all reporting groups
Arm/Group | High ACE Activity Fresh Frozen Plasma | Normal Saline | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] |  | 47.9 [37.1 to 58.1] | 47.9 [37.1 to 58.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 2 | 2
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Determine if Treatment With 2 Units of Fresh Frozen Plasma That Contains ≥ 50 U/L of ACE Activity Increases Serum ACE Activity
Description: The subjects' serum ACE activity will be assessed prior to treatment and 30 minutes after treatment and compared to determine if the treatment increases serum ACE activity
Time Frame: Compare serum ACE activity before treatment and 30 minutes after treatment
Population: Blood was never drawn due to pandemic related issues, the subjects' serum ACE activity were not assessed/drawn prior to treatment and nor 30 minutes after treatment, no result data available.
Arm/Group | High ACE Activity Fresh Frozen Plasma | Normal Saline
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Determine How Treatment Affects the Severity of Angioedema Using a Published Validated Clinical Rating Scale
Description: The severity of the the subjects' angioedema will be assessed using a published validated clinical rating scale before treatment and at 30 minutes, 2 hours, and 8 hours after treatment
Time Frame: Compare angioedema severity before treatment and 30 minutes, 2 hours, and 8 hours after treatment
Population: Due to pandemic related issues, no data was collected. Clinical rating scale was never done.
Arm/Group | High ACE Activity Fresh Frozen Plasma | Normal Saline
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Sustained Change in Serum ACE Activity With Treatment
Description: Determine if treatment results in a sustained change in ACE activity levels
Time Frame: Compare serum ACE activity before treatment and at 2 hours and 8 hours after treatment
Population: Due to pandemic related issues,sustained change in serum ACE activity with treatment was never collected.
Arm/Group | High ACE Activity Fresh Frozen Plasma | Normal Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients were observed for adverse effects during their ED visit only, or up to 24 hours. No further monitoring was conducted after the patient was discharged from the ED. Both participants received placebo (normal saline).
Description: Both enrolled participant were randomized to the placebo arm, which they recieved normal saline..
Arm/Group | High ACE Activity Fresh Frozen Plasma | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT04679311/Prot_SAP_000.pdf